CLINICAL TRIAL: NCT02052661
Title: Persistence of Hepatitis B Antibodies, Immunogenicity and Safety of GSK Biologicals' Hepatitis B Vaccine Engerix™-B Kinder (SKF103860) Challenge Dose in Adolescents Vaccinated With Four Doses of Infanrix™ Hexa (SB217744) During Infancy
Brief Title: This Study Aims to Determine the Long-term Persistence of Antibodies Against Hepatitis B and to Evaluate the Immunogenicity and Safety of Hepatitis B Vaccine in Adolescents Vaccinated in Infancy With Infanrix™ Hexa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 106793; 2013-002821-41 (EudraCT Number)
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Results first posted 2015-08-27 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2017-04

CONDITIONS: Hepatitis B
Keywords: Infanrix™ hexa; Hepatitis B antibodies; Immunogenicity; Hepatitis B; Adolescents; Infancy; Engerix™-B Kinder; Safety
MeSH Terms: conditions — Hepatitis B

ARMS (1):
- Engerix-B Kinder Group (Experimental): Subjects who were previously primed and boosted with four doses of Infanrix™ hexa in the first two years of life, received a single dose of Engerix™-B Kinder vaccine. The vaccine was administered intramuscularly into the deltoid of the non-dominant arm.
  Interventions: Biological: Engerix™-B Kinder

INTERVENTIONS:
Biological: Engerix™-B Kinder — Single dose administered intramuscularly in deltoid region of non-dominant arm.

SUMMARY:
The purpose of this study is to assess the long-term persistence of immunity to hepatitis B in adolescents aged 12-13 years who were vaccinated with four doses of Infanrix™-Hexa in infancy and to assess the anamnestic response, immunogenicity, safety and reactogenicity of a single challenge dose of the hepatitis B vaccine Engerix™-B Kinder.

ELIGIBILITY:
Inclusion Criteria:

* Subjects' parent(s)/LAR(s) who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g. completion of the diary cards, return for follow-up visit).
* A male or female between the ages of 12 to 13 (from and including the 12th birthday, up to but excluding the 14th birthday) at the time of enrolment.
* Subjects with documented evidence of previous vaccination with four consecutive doses of Infanrix hexa as part of routine vaccination in Germany: three doses of primary vaccination received by 9 months of age and one booster dose received between 11 and 18 months of age.
* Written informed consent obtained from the parents/LAR(s) of the subject.

  * In addition to the informed consent that will be signed by the parents/LAR(s), written informed assent of the subject will be sought.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Administration of long-acting immune-modifying drugs at any time during the study period (e.g. infliximab).
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs within six months prior to the vaccination. Inhaled and topical steroids are allowed.
* Administration of any chronic drug therapy to be continued during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before and ending 30 days after the HBV challenge dose, with the exception of tetanus toxoid, reduced diphtheria toxoid and acellular pertussis (dTpa) vaccine, which can be given as part of routine vaccination practice.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product (pharmaceutical product or device).
* Evidence of previous hepatitis B booster vaccination since administration of the fourth dose of Infanrix hexa booster in the second year of life.
* History of or intercurrent hepatitis B disease.
* Hepatitis B vaccination at birth.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness including thrombocytopenia and bleeding disorders.
* History of any neurological disorders or seizures.
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥ 37.5°C for oral, axillary or tympanic route, or ≥ 38.0°C on rectal route. The preferred route for recording temperature in this study will be axillary.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may, be enrolled at the discretion of the investigator.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the dose of study vaccine or planned administration during the study period.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Ages: 12 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 301 (Actual)
Dates: Start 2014-02-18; Primary Completion 2014-09-23 (Actual); Study Completion 2014-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- Germany (11):
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Tuttlingen, Baden-Wurttemberg
  - GSK Investigational Site, Bindlach, Bavaria
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Löhne, North Rhine-Westphalia
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Radebeul, Saxony
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Neumünster

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 106793 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 106793 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106793 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106793 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106793 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106793 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106793 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 301 subjects were enrolled in the study but one subject was withdrawn before any study procedure.
Groups:
- Engerix-B Kinder Group: Subjects who were previously primed and boosted with four doses of Infanrix hexa in the first two years of life, received a single dose of Engerix-B Kinder vaccine. The vaccine was administered intramuscularly into the deltoid of the non-dominant arm.
Period: Overall Study
Arm/Group | Engerix-B Kinder Group
Started | 300
Completed | 300
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 300
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.3 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150
  Male | 150

OUTCOME MEASURES:

1. Primary Outcome: Anti-HBs Immune Response
Description: Anti-HBs immune response was defined as the number of subjects with Anti-HBs antibody concentrations ≥ 100 mIU/ml.
Time Frame: One month after the single challenge dose of Engerix-B Kinder vaccine (Month 1)
Population: The analysis was performed on the According-To-Protocol cohort for immunogenicity, which included all evaluable subjects, who complied with the protocol, for whom immunogenicity data were available and for whom assay results were available for antibodies against at least one study vaccine antigen component at the post-vaccination time points.
Measure: Number; unit: Subject
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 289
Subject | 272

2. Secondary Outcome: Anti-HBs Antibody Concentrations at 12-13 Years of Age, After Previous Vaccination With Infanrix Hexa.
Description: Concentrations were expressed as geometric mean concentrations (GMCs) for the seropositivity cut-off of 6.2 mIU/ml.
Time Frame: Before (PRE) and 1 month after (POST) the single challenge dose of Engerix-B Kinder vaccine.
Population: The analysis was performed on the According-To-Protocol cohort for persistence, which included all evaluable subjects, aged 12-13 years at the time of enrolment, who did not received any additional dose of hepatitis B vaccine other than four doses of Infanrix hexa during first two years of life, for whom the serological results were available.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 293
mIU/mL
  Anti-HBs, PRE: number analyzed (Participants) | 291
  Anti-HBs, PRE | 22.7 [18.5 to 27.9]
  Anti-HBs, POST: number analyzed (Participants) | 289
  Anti-HBs, POST | 3502.6 [2672 to 4591.5]

3. Secondary Outcome: Number of Subjects With Anti-HBs Antibody Concentrations ≥ 6.2 mIU/ml, ≥ 10 mIU/ml, 10 to < 100 mIU/ml and ≥ 100 mIU/ml.
Description: A seropositive subject was defined as a subject with anti-HBs antibody concentrations ≥ 6.2 milli-international units per milliliter (mIU/ml). A seroprotected subjects was defined as a subject with anti-HBs antibody concentrations ≥ 10 mIU/ml.
Time Frame: Before the single challenge dose of Engerix-B Kinder vaccine.
Population: as for outcome 2
Measure: Number; unit: Subject
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 293
Subject
  Anti-HBs ≥ 6.2 mIU/ml | 205
  Anti-HBs ≥ 10 mIU/ml | 178
  Anti-HBs 10 to < 100 mIU/ml | 116
  Anti-HBs ≥ 100 mIU/ml | 62

4. Secondary Outcome: Number of Subjects With Anti-HBs Antibody Concentrations ≥ 6.2 mIU/ml and ≥ 10 mIU/ml.
Description: A seropositive subject was defined as a subject with anti-HBs antibody concentrations ≥ 6.2 mIU/ml. A seroprotected subjects was defined as a subject with anti-HBs antibody concentrations ≥ 10 mIU/ml.
Time Frame: 1 month after the single challenge dose of Engerix-B Kinder vaccine.
Population: as for outcome 1
Measure: Number; unit: Subject
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 289
Subject
  Anti-HBs ≥ 6.2 mIU/ml | 283
  Anti-HBs ≥ 10 mIU/ml | 282

5. Secondary Outcome: Number of Subjects With an Anamnestic Response to the Single Challenge Dose of Engerix-B Kinder Vaccine.
Description: The amnestic response to the challenge dose was defined as: for initially seronegative subjects, antibody concentration ≥ 10mIU/mL; for initially seropositive subjects, antibody concentration at least four times the pre-challenge antibody concentration.
Time Frame: One month after the single challenge dose of Engerix-B Kinder vaccine.
Population: as for outcome 1
Measure: Number; unit: Subject
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 287
Subject | 277

6. Secondary Outcome: Number of Subjects With Any Solicited Local Symptoms.
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 4-day (Day 0-3) follow-up period after the single challenge dose of Engerix-B Kinder vaccine.
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with the vaccine administration documented.
Measure: Number; unit: Subject
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 300
Subject
  Pain | 132
  Redness | 70
  Swelling | 29

7. Secondary Outcome: Number of Subjects With Any Solicited General Symptoms.
Description: Assessed solicited general symptoms were fatigue, gastrointestinal, headache and temperature [defined as axillary temperature equal to oe above 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 4-day (Day 0-3) follow-up period after the single challenge dose of Engerix-B Kinder vaccine.
Population: as for outcome 6
Measure: Number; unit: Subject
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 300
Subject
  Fatigue | 73
  Gastrointestinal | 34
  Headache | 71
  Temperature/(Axillary) | 7

8. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs).
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Day 0-30) follow-up period after the single challenge dose of Engerix-B Kinder vaccine.
Population: as for outcome 6
Measure: Number; unit: Subject
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 300
Subject | 44

9. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs).
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Month 0 to Month 1
Population: as for outcome 6
Measure: Number; unit: Subject
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 300
Subject | 2

ADVERSE EVENTS:
Time Frame: Solicited symptoms: during the 4-day (Day 0-3) follow-up period after vaccination Unsolicited AEs: during the 31-day (Day 0-30) follow-up period after vaccination SAEs: During the entire study.
Description: The occurrence of reported AEs (all/related) was not available and is encoded as equal to the number of subjects affected.
Arm/Group | Engerix-B Kinder Group
Serious Adverse Events (participants affected / at risk) | 2/300
Other Adverse Events (participants affected / at risk) | 200/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Engerix-B Kinder Group (N=300)
Contusion (Injury, poisoning and procedural complications) | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Engerix-B Kinder Group (N=300)
Pain (General disorders) | 132
Redness (General disorders) | 70
Swelling (General disorders) | 29
Fatigue (General disorders) | 73
Gastrointestinal (General disorders) | 34
Headache (General disorders) | 71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.